CLINICAL TRIAL: NCT06142110
Title: Investigation of The Relationship Between Functional Movement and Respiratory Muscle Strength in Professional Football Players and Sedentary Individuals: A Controlled Trial
Brief Title: The Relationship Between Functional Movement and Respiratory Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Research assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMS and RMS
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Functional Movement Quality; Respiratory Muscle Strength; Core Stability; Injury
Keywords: Functional movement; Respiratory muscle; core; injury; sports
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A controlled trial was conducted by including all professional football players in the city and an equivalent number of sedentary individuals
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment of professional football player (Active Comparator): Respiratory muscle strength and functional movement quality of professional football players were evaluated. Functional movement screen and portable spirometer were used for evaluation.
  Interventions: Other: Funcional movement screen; Diagnostic Test: Respiratory muscle strength
- Assessment of sedantery individuals (Active Comparator): Respiratory muscle strength and functional movement quality of sedantery individuals were evaluated. Functional movement screen and portable spirometer were used for evaluation.
  Interventions: Other: Funcional movement screen; Diagnostic Test: Respiratory muscle strength

INTERVENTIONS:
Other: Funcional movement screen — FMS is a biomechanical screening and evaluation method to reveal the limitations and asymmetries on the 7 basic movement patterns, which are the determinants of functional movement quality.
Diagnostic Test: Respiratory muscle strength — Respiratory muscle strength was assessed with an additional mouthpiece attached to the portable spirometer as maximum inspiratory pressure and maximum expiratory pressure.

SUMMARY:
Functional Movement Screen (FMS) is a battery used for injury prediction, identifying asymmetry and weak connections in basic functional movement patterns. The muscles assessed in FMS are also respiratory muscles. Therefore, FMS scores were thought to be related to respiratory muscle strength. The aim of our study was to examine the relationship between Functional Movement Screen and respiratory muscles strength in professional football players and sedentary individuals.

DETAILED DESCRIPTION:
Predicting and preventing sports injuries is very important for football players to maintain high performance. The measurement methods used to predict the injury probabilities of football players are quite expensive. However, in recent years, the Functional Movement Screen (FMS), used as an injury estimation tool in football players, can be easily applied in the field without the need for expensive equipment.

FMS is a biomechanical screening and evaluation method to reveal the limitations and asymmetries on the 7 basic movement patterns, which are the determinants of functional movement quality. FMS test battery aims to evaluate movements that require muscle strength, flexibility, range of motion, coordination, balance and proprioception. In the test; joint range of motion, asymmetry of motion, trunk strength and stabilization, balance, neuromuscular coordination, flexibility and dynamic flexibility properties are determined in a non-invasive, easy and economical way. Spine and core stabilization skills are exhibited in the movements included in the FMS.

In the literature, there is no study examining the relationship between respiratory muscle strength and FMS in football players and healthy individuals. However, respiratory mechanics play an important role in posture and spine stabilization have been shown.

Many functional activities in sports require trunk stabilization to transfer force symmetrically between the extremities. Impaired postural control, poor balance, lack of proprioception, and poor motor control have been shown to cause pain and disability and interfere with normal movement . Primary or accessory respiratory muscles; diaphragm, intercostal muscles, serratus anterior and posterior, pectorals, abdominal wall muscles also contribute to core and body stabilization. Therefore, it was thought that there may be a relationship between inspiratory and expiratory muscle strength and the quality of movements requiring trunk stabilization, balance and symmetry. In order to reveal this relationship, it is necessary to examine the relationship between FMS scores and respiratory muscle strength of trained/untrained individuals with different body types and movement patterns. Based on these assumptions, this study aimed to examine the FMS scores and respiratory muscles strength to investigate relationship between functional movement quality and respiratory muscles in professional football players and sedentary individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy professional football players, healthy sedantery individuals

Exclusion Criteria:

* Subject with Cardiovascular, respiratory disease, inflammatory disease, smokers and acute injury

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Functional movement Screen | from enrollment to the end of assessment for 1 day
  FMS was designed to identify asymmetries, limitations and compensations of the football players throughout the movement pattern, not in the joints. It consists of seven basic movements; Deep squad, hurdle steps, inline lunge, shoulder mobility, active straight leg rise, trunk stability push up, and rotator stability. The FMS tests are scored on a scale of 0 to 3, with the sum creating a composite score ranging from 0 to 21 points. Higher scores mean better conditions
Respiratory muscle strength | from enrollment to the end of assessment for 1 day
  Respiratory muscle strength is evaluated by individuals performing maximal expiration and inspiratory maneuvers.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ünver, Professor, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No